CLINICAL TRIAL: NCT00001031
Title: A Phase II Clinical Trial to Evaluate the Immunogenicity and Reactogenicity of the Recombinant HIV-1 Envelope Vaccines SF-2 rgp120 (CHO) [Chiron Vaccines] in MF59 Adjuvant and MN rgp120/HIV-1 [VaxGen] in Alum Adjuvant in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biocine (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 201; 10588 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: rgp120/HIV-1MN
Biological: rgp120/HIV-1 SF-2

SUMMARY:
To evaluate the safety and immunogenicity of SF-2 rgp120 vaccine in MF59 versus MN rgp120 vaccine in alum in volunteers who are seronegative for HIV-1. AS PER AMENDMENT 07/02/97: To determine the ability of immunization with MN rgp120/HIV-1 in combination with alum or SF-2 rgp120 in combination with MF59 to induce an HIV-1 envelope-specific delayed-type hypersensitivity (DTH) response in volunteers who receive rsgp120/MN skin testing.

The amino acid sequence of HIV-1 gp120 can vary as much as 40 percent from isolate to isolate. Thus, the identification of an immunogen that can elicit broadly neutralizing antibodies to HIV-1 is a major challenge in AIDS vaccine development. Two candidate vaccines, recombinant envelope subunit proteins from the SF-2 and MN isolates of HIV-1, have shown immunogenicity and good tolerance in healthy immunocompetent adults. This study will expand testing into a larger population base, particularly targeting individuals at high risk for HIV infection.

DETAILED DESCRIPTION:
The amino acid sequence of HIV-1 gp120 can vary as much as 40 percent from isolate to isolate. Thus, the identification of an immunogen that can elicit broadly neutralizing antibodies to HIV-1 is a major challenge in AIDS vaccine development. Two candidate vaccines, recombinant envelope subunit proteins from the SF-2 and MN isolates of HIV-1, have shown immunogenicity and good tolerance in healthy immunocompetent adults. This study will expand testing into a larger population base, particularly targeting individuals at high risk for HIV infection.

HIV-seronegative volunteers (including four populations at higher risk for HIV infection and two populations at lower risk) receive one of four regimens. Two treatment groups receive 50 mcg SF-2 rgp 120 (BIOCINE) in MF59 adjuvant or 600 mcg MN rgp120 (Genentech) in alum. Two control groups receive vehicle (placebo) in MF59 adjuvant alone or alum adjuvant alone. Immunizations are given at months 0, 1, and 6. AS PER AMENDMENT 10/93: patients enrolled by June 15, 1993, receive a fourth immunization at month 12 or 18 (50 percent of patients for each schedule). Patients are followed until 2 years after the first injection. AS PER AMENDMENT 05/10/94: a special study of vaccine acceptability and HIV-related risk behavior will be conducted at some time between months 12 and 18. AS PER AMENDMENT 07/02/97: a special DTH study will be conducted in consenting volunteers who have received three or four immunizations. The injections will be given at the end of the study (on or after day 1, & 56). Followup is extended to 56 days after administration of the intradermal injection.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* HIV negativity by ELISA.
* CD4 count >= 400 cells/mm3.
* No clinically significant medical disease.
* No history of immunodeficiency, autoimmune disease, or use of immunosuppressive medication.
* No prior HIV vaccines.
* Classification in one of the eligible risk groups defined in the Disease Status field.

Eligible higher risk groups:

* Heterosexual teenagers and young adults (ages 16-28 permitted) who have attended a clinic for sexually transmitted diseases in the last 3 months or have higher risk sexual behavior.
* Homosexually active males who are practicing higher risk behavior (ages 18-60).
* Injection drug users active within the past 3 years (ages 18-60).
* Heterosexual partners of HIV seropositive individuals (ages 18-60).

Eligible lower risk groups:

* Homosexually active males who are practicing lower risk behavior (ages 18-60).
* Adult women and heterosexual adult men practicing lower risk sexual behavior (ages 18-60).

Exclusion Criteria

Prior Medication:

Excluded:

* Prior HIV vaccines.
* Prior immunosuppressive medications.
* Experimental agents within the past 30 days.
* AS PER AMENDMENT 07/02/97: Use of systemic steroids in the past month (for volunteers undergoing DTH testing).

AS PER AMENDMENT 07/02/97:

* History of eczema or allergic-type reactions to vaccines used in protocol 201 (for volunteers undergoing DTH testing).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 296 (Actual)
Dates: Study Completion 1997-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair; McElrath J, Study Chair
Locations (7):
- United States (7):
  - UAB AVEG, Birmingham, Alabama
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - JHU AVEG, Pittsburgh, Pennsylvania
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] McElrath MJ, Corey L, Clements ML, Belshe R, Keefer M, Graham B, Fast P, Matthews T, Duliege AM, Francis D. A phase II HIV vaccine trial in seronegative subjects: safety, immunogenicity, and future directions. Int Conf AIDS. 1994 Aug 7-12;10(1):91 (abstract no 317A)
- [Background] McElrath MJ, Montefiori DM, Clements ML, Belshe RB, Dolin R, Graham BS, Duliege A-M, Francis D, Bolognesi DP, Matthews TJ, Wolff M, Fast P, Corey L. Longitudinal vaccine-induced immunity and risk behavior of study participants of AVEG phase II protocol 201. Conf Adv AIDS Vaccine Dev. 1996 Feb 11-15;216 [Poster 96]
- [Background] McElrath MJ, Corey L, Montefiori D, Wolff M, Schwartz D, Keefer M, Belshe R, Graham BS, Matthews T, Wright P, Gorse G, Dolin R, Berman P, Francis D, Duliege AM, Bolognesi D, Stablein D, Ketter N, Fast P. A phase II study of two HIV type 1 envelope vaccines, comparing their immunogenicity in populations at risk for acquiring HIV type 1 infection. AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 2000 Jun 10;16(9):907-19. doi: 10.1089/08892220050042846. PMID 10875616
- [Background] Harrison K, Vlahov D, Jones K, Charron K, Clements ML. Medical eligibility, comprehension of the consent process, and retention of injection drug users recruited for an HIV vaccine trial. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Nov 1;10(3):386-90. PMID 7552502
- [Background] McElrath MJ, Montefiori D, Wolff M, Clements M, Gorse G, Keefer M, Graham B, Duliege AM, Francis D, Matthews T, Fast P, Corey L. Safety, immunity, and risk behavior in HIV-1-uninfected volunteers representing diverse risk populations following recombinant envelope vaccinations: a three-year followup. Int Conf AIDS. 1996 Jul 7-12;11(1):10 (abstract no MoA284)